CLINICAL TRIAL: NCT01323049
Title: Comparison of Spontaneous Ventilation Time in Air Without Desaturation After Positive Pressure Extubation Versus Aspiration Extubation When Awakening From General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2010/JL-03; 2011-A00051-40 (Other: ANSM)
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Anesthesia, General
Keywords: extubation strategy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive pressure extubation (Active Comparator): Positive pressure extubation will be used for patients waking up from general anesthesia in this group
  Interventions: Procedure: Positive pressure extubation
- Aspiration/suction extubation (Active Comparator): Aspiration/suction extubation will be used for patients waking up from general anesthesia in this group
  Interventions: Procedure: Aspiration/suction extubation

INTERVENTIONS:
Procedure: Positive pressure extubation — Positive pressure extubation will be used for patients waking up from general anesthesia
  Arms: Positive pressure extubation
Procedure: Aspiration/suction extubation — Aspiration/suction extubation will be used for patients waking up from general anesthesia
  Arms: Aspiration/suction extubation

SUMMARY:
The primary objective is to show that positive pressure extubation improves oxygenation immediately after extubation compared to extubation via "aspiration" by evaluating and comparing the onset time of desaturation during spontaneous ventilation during awakening following general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 1 hour of follow up
* ASA 1 to 3
* The patient is schedules for orthopedic surgery (limbs) with general anesthesia

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* The patient is breastfeeding
* Chronic respiratory insufficiency
* Cardiopathy
* Obstructive sleep apnea
* Two or more predictive criteria for difficult mask ventilation (age > 55 years, toothless, beard, snorer, BMI > 26)
* No predictive criteria for difficult intubation (SPIDS <= 10)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02-25 (Actual); Study Completion 2014-02-25 (Actual)

PRIMARY OUTCOMES:
Spontaneous ventilation (air) time without desaturation after extubation (min) | 10 minutes
  desaturation is defined as an SpO2< 92%

SECONDARY OUTCOMES:
presence/absence of a desaturation after extubation | 10 minutes
  desaturation is defined as an SpO2<92%
minimum Sp02 level after extubation (%) | 10 minutes
minimum Sp02 level after extubation (%) | 60 minutes
presence/absence of complications | 60 minutes
  coughing, airway obstruction, laryngospasm, desaturation, apnea, vomiting in the first hour
presence / absence of therapeutic maneuvers | 60 minutes
  includes oxygen therapy (or bezel ventimasque), Guedel airway, mask assistance, re-intubation during the first hour
presence/absence of any complication | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joël L'Hermite, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France

REFERENCES:
- [Result] L'Hermite J, Wira O, Castelli C, de La Coussaye JE, Ripart J, Cuvillon P. Tracheal extubation with suction vs. positive pressure during emergence from general anaesthesia in adults: A randomised controlled trial. Anaesth Crit Care Pain Med. 2018 Apr;37(2):147-153. doi: 10.1016/j.accpm.2017.07.005. Epub 2017 Sep 4. PMID 28882741